CLINICAL TRIAL: NCT04507139
Title: Early Longitudinal Imaging in Parkinson's Progression Markers Initiative Using [¹⁸F] AV-133 and DaTscan™ (PPMI Early Imaging)
Brief Title: Early Longitudinal Imaging in Parkinson's Progression Markers Initiative Using [¹⁸F] AV-133 and DaTscan™
Status: Active, not recruiting | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Ken Marek, MD, Protocol Principal Investigator, Institute for Neurodegenerative Disorders
Other Study IDs: PPMI-004
Record Dates: First submitted 2020-08-03; First posted 2020-08-11 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Bio-markers; Neurodegenerative disorder; Imaging; Prodromal; Genetics; At Risk; Loss of Smell
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Anosmia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Directly examine whether early (6-month) imaging with DaTscan and [¹⁸F] AV-133 will provide an early signal of disease progression in recently diagnosed untreated PD patients.

DETAILED DESCRIPTION:
The study is a longitudinal, multi-center study to assess progression of DaTscan and [18F] AV-133 imaging in PD and Prodromal patients. Participants will be followed for up to 24 months. Approximately 50 early PD participants and 100 Prodromal participants will be recruited from up to 15 sites. Participants will be comprehensively assessed at baseline and follow up according to the Schedule of Activities for the respective cohort. Participants will undergo imaging assessments with DaTscan and [18F] AV-133 and clinical (motor, neuropsychiatric and cognitive) assessments. Data will be collected by each site under uniformly established protocols and data will be stored and analyzed at designated core facilities.

ELIGIBILITY:
Inclusion Criteria:

1. A PD participant consented to PPMI Clinical, or, a Prodromal participant confirmed eligible to proceed to PPMI Clinical Baseline visit.
2. Able to provide informed consent.
3. Women may not be pregnant, lactating or planning pregnancy during the study.

   * Includes a negative serum pregnancy test prior to Baseline 18F-AV-133 injection.
   * Includes a negative urine pregnancy test prior to injection of 18F-AV-133 on day of Baseline PET scan.
   * Women participating in the study must be of non-childbearing potential or be using a highly effective method of birth control 14 days prior to until at least 24 hours after the last injection of 18F-AV-133.

     * Non-childbearing potential is defined as a female that must be either postmenopausal (no menses for at least 12 months prior to Screening) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy).
     * Highly effective method of birth control is defined as practicing at least one of the following: A birth control method that results in a less than 1% per year failure rate when used consistently and correctly, such as oral contraceptives for at least 3 months prior to injection, an intrauterine device (IUD) for at least 2 months prior to injection, or barrier methods, e.g., diaphragm or combination condom and spermicide. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.

Exclusion Criteria:

1. Received any of the following medications that might interfere with 18F- AV-133 PET imaging: tetrabenazine (TBZ) or methylphenidate, reserpine, or amphetamine derivative, within 1 month prior to the Baseline 18F-AV-133 injection.
2. Have current clinically significant cardiovascular disease or abnormalities on screening ECG (including but not limited to QTc > 450 msec).
3. Are currently taking medications that are known to cause QT- prolongation
4. Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 early PD and 100 prodromal participants will be recruited from up to 15 sites internationally.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Mean Rate of Change | 24 months
  The mean rates of change and the variability around the mean of imaging outcomes in early and Prodromal PD patients, and where appropriate the comparison of these rates between PD patient subsets at study intervals ranging from 6 months to 24 months. Specific examples of outcomes include dopamine transporter striatal uptake and vesicular monoamine transporter type-2 uptake. PD patient subsets may be defined by baseline assessments, genetic mutation, progression milestones and/or rate of clinical, imaging, or biomic change.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Institute For Neurodegenerative Disorders, New Haven, Connecticut
  - Boston University Medical Center, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania